CLINICAL TRIAL: NCT06475742
Title: A Phase 3, Multicenter, Open-label, Single-arm, Extension Study to Evaluate the Long-term Safety and Tolerability of Cenerimod in Adult Subjects With Moderate-to-Severe Systemic Lupus Erythematosus (SLE) on Top of Background Therapy
Brief Title: Long-term Safety and Tolerability of Cenerimod in Adults With Systemic Lupus Erythematosus
Acronym: OPUS OLE
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID-064A303; 2024-514354-67-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-08

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Skin and Connective Tissue Diseases; Connective Tissue Diseases; Immune System Diseases; Autoimmune Diseases; Musculoskeletal and connective tissue disorders
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Skin and Connective Tissue Diseases; Connective Tissue Diseases; Immune System Diseases; Autoimmune Diseases | interventions — cenerimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cenerimod 4 mg (Experimental): Participants will receive oral cenerimod once daily in addition to background systemic lupus erythematosus therapy, for at least 1 year and up to a maximum of 3 years.
  Interventions: Drug: Cenerimod

INTERVENTIONS:
Drug: Cenerimod — Film-coated tablets at a dose of 4 mg.
  Other Names: ACT-334441

SUMMARY:
The goal of this clinical study is to learn about the long-term safety and tolerability of cenerimod in adult patients with moderate to severe symptoms of systemic lupus erythematosus.

The main questions it aims to answer are:

* Whether cenerimod causes any adverse effects ('side effects') when given on top of drugs already being given for systemic lupus erythematosus.
* How well cenerimod works to reduce symptoms of systemic lupus erythematosus when taken for at least 1 year and up to 3 years.

Participants taking part in this study will have already taken part in another study, where they received either cenerimod or placebo (look-alike substance containing no active drug) for 1 year.

In this clinical study approximately 680 participants will receive cenerimod (on top of drugs already being given for systemic lupus erythematosus) for at least 1 year and up to 3 years.

DETAILED DESCRIPTION:
Participants who completed the 12-month double-blind treatment period (cenerimod 4 mg or placebo) in either of the parent studies, ID-064A301 or ID-064A302, are eligible to participate in this extension study.

All participants in this study will receive cenerimod 4 mg for at least 12 months (1 year) and up to a maximum of 36 months (3 years). All participants may additionally receive standard of care treatment for systemic lupus erythematosus, i.e., at least 1 of the following: oral corticosteroids, antimalarial drugs, or immunosuppressant drugs.

When all participants have reached at least 12 months of study treatment or have prematurely discontinued study treatment before the end of Month 12, the end-of-treatment will be scheduled for all participants who are still on study treatment.

The safety follow-up period starts on the day after the last dose of study treatment and ends after 6 months with the final study visit. Thus, the maximum duration of participation is 3.5 years.

Data collected in this extension study will allow an assessment of whether the safety and tolerability profile of cenerimod established in the controlled parent studies remains the same after a longer period of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form prior to any study-mandated procedure.
2. Participants with a diagnosis of systemic lupus erythematosus who:

   * Completed the 12-month double-blind treatment period of either of the parent studies (ID-064A301, ID-064A302).
   * Did not meet any study treatment stopping criteria during the parent study.
   * Completed the last scheduled visit of the parent study. Participants who did not complete the last scheduled visit for reasons beyond their control may be eligible for this study upon approval by the sponsor.
3. Women of child-bearing potential:

   * Negative pregnancy test at Visit 1.
   * Agreement to undertake monthly urine pregnancy tests from Visit 2 up to 6 months after study treatment discontinuation.
   * Agreement to use a highly effective method of contraception from Visit 1 up to 6 months after study treatment discontinuation.

Exclusion Criteria:

1. Poor compliance with study-mandated procedures during the parent study (ID-064A301 or ID-064A302), e.g., took less than 80% of the planned doses of double-blind study treatment; or did not attend a majority of the site visits, unless there was a medically justified reason as judged by the investigator.
2. Systemic lupus erythematosus driven renal disease, central nervous system lupus, or active severe or unstable neuropsychiatric systemic lupus erythematosus where, in the judgment of the investigator, protocol-specific systemic lupus erythematosus background therapy is insufficient, and the use of a more aggressive therapeutic approach or other treatments not permitted in the protocol is indicated.
3. Women of child-bearing potential planning to become pregnant up to the final study visit.
4. Judged not eligible to participate by the investigator, for any other reason.
5. Confirmed active or latent tuberculosis (applicable only if requested by local regulations).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | Day 1 (post dose) to a maximum of 3.5 years
  Occurrence of treatment-emergent adverse events up to the final study visit (maximum 3 years of study treatment plus 6-month safety follow-up period).
Serious adverse events | Day 1 (post dose) to a maximum of 3.5 years
  Occurrence of serious adverse events up to the final study visit (maximum 3 years of study treatment plus 6-month safety follow-up period).
Adverse events of special interest | Day 1 (post dose) to a maximum of 3.5 years
  Occurrence of adverse events of special interest up to the final study visit (maximum 3 years of study treatment plus 6-month safety follow-up period).
  Adverse events of special interest include the anticipated risks of treatment with cenerimod, known class effects, and events that may be related to systemic lupus erythematosus comorbidities, i.e., adverse events related to:
  * Effects on heart rate and rhythm
  * Hypotension
  * Hypertension
  * Cardiovascular
  * Hepatobiliary disorders / liver enzyme abnormalities
  * Pulmonary
  * Eye disorders
  * Infections
  * Skin malignancies
  * Non-skin malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (85):
- United States (10):
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Omega Research MetroWest, LLC, DeBary, Florida
  - SouthCoast Research Center, Inc., Miami, Florida
  - D&H National Research Centers INC, Miami, Florida
  - San Marcus Res Clin Inc., Miami Lakes, Florida
  - Accurate Clinical Research Inc. - Lake Charles, Lake Charles, Louisiana
  - RB Wellness Clinic, Las Vegas, Nevada
  - Accurate Clinical Research Inc - (Najam), Baytown, Texas
  - Novel Research LLC, Bellaire, Texas
  - Accurate Clinical Research Inc., Houston, Texas
- Argentina (8):
  - Aprillus Asistencia e Investigacion, Buenos Aires
  - Centro Médico Arsema, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - IR Medical Center S.A., Mendoza
  - Instituto Medico CER, Quilmes
  - Instituto CAICI SRL, Rosario
  - Centro de investigaciones medicas Tucuman, San Miguel de Tucumán
  - ICT (Investigaciones Clínicas Tucumán), San Miguel de Tucumán
- LMK Servicos Medico S/S, Porto Alegre, Brazil
- Bulgaria (2):
  - Outpatient Clinic for Specialized Outpatient Medical Care - Medical Center Kyuchuk Parizh Ltd., Plovdiv
  - DCC Equita EOOD, Varna
- Chile (6):
  - Enroll SpA, Providencia
  - Biomedica Research Group, Providencia
  - Sociedad Médica del Aparato Locomotor S. A., Providencia
  - Centro de Especialidades Medicas Vanguardia, Temuco
  - Clinical Research Chile SpA, Valdivia
  - Hospital San José de Victoria, Victoria
- Czechia (2):
  - iMedica s.r.o., Brno
  - Institute of Rheumatology Prague, Prague
- Georgia (11):
  - LTD "New Plasma Clinic", Batumi
  - Institute of Clinical Cardiology, Ltd, Tbilisi
  - LTD "Tbilisi Central Hospital", Tbilisi
  - National Institute of Endocrinology Ltd., Tbilisi
  - Tbilisi Heart and Vascular Clinic Ltd., Tbilisi
  - Aversi Clinic LTD, Tbilisi
  - Medi Club Georgia Ltd., Tbilisi
  - Ltd. Mtskheta Street Clinic, Tbilisi
  - The First Medical Center Ltd., Tbilisi
  - LLC "Innova", Tbilisi
  - LTD "Tbilisi Heart Center", Tbilisi
- Germany (2):
  - Universitatsklinikum Leipzig, Leipzig
  - Klinik für Rheumatologie und Klinische Immunologie, Minden
- Greece (4):
  - General Hospital of Athens "Hippokration", Athens
  - Euromedica - Kyanos Stavros, Thessaloniki
  - General Hospital of Thessaloniki "Hippokration", Thessaloniki
  - 424 General Military Hospital, Thessaloniki
- Peru (3):
  - Centro de Investigación del Hospital Militar Central, Jesus Maria
  - Unidad de Investigación de la Clinica International, San Borja
  - Investigaciones Clinicas / Instituto de Ginecologa y Reproduccion, Santiago de Surco
- Philippines (8):
  - Chong-Hua Hospital, Cebu City
  - Lipa Medix Medical Center, Lipa City
  - Makati Medical Center, Makati
  - Ospital ng Makati, Makati
  - St Lukes Medical Center, Quezon City
  - Far Eastern University - Nicanor Reyes Medical Foundation, Quezon City
  - St Luke's Medical Center Quezon City / University of Santo Tomas Hospital, Sampaloc
  - Jose R. Reyes Memorial Medical Center, Santa Cruz
- Poland (7):
  - Szpital Uniwersytecki nr 2 im. dr. Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Medyczne Pratia Częstochowa, Częstochowa
  - Centrum Medyczne Angelius Provita, Katowice
  - Vita Longa Sp. z o.o., Katowice
  - Medyczne Centrum Hetmanska, Poznan
  - Twoja Przychodnia Poznańskie Centrum Medyczne, Poznan
  - Malwa-Med Iwona Chlebicka, Wroclaw
- Portugal (5):
  - Hospital Prof. Doutor Fernando Fonseca, Amadora
  - Centro Hospitalar Universitário do Algarve - Hospital de Faro, Faro
  - ULS Guarda, Guarda
  - Hospital Senhora Oliveira-Guimaraes, Guimarães
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E., Vila Nova de Gaia
- Puerto Rico (2):
  - Centro Reumatologico de Caguas, Caguas
  - GCM Medical Group, PSC, San Juan
- Centrul Medical de Diagnostic si Tratament Ambulatoriu Neomed S.R.L, Brasov, Romania
- Serbia (3):
  - Institute of Rheumatology, Belgrade, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - Special Hospital for Rheumatic Diseases, Novi Sad, Novi Sad
- South Africa (2):
  - Panorama Medical Centre, Panorama
  - Charlotte Maxeke Johannesburg Academic Hospital, Parktown
- Seoul National University Hospital, Seoul, South Korea
- Spain (4):
  - Parc Taulí Sabadell University Hospital, Sabadell
  - Clinica Gaias Santiago, Santiago de Compostela
  - Hospital QuironSalud Sagrado Corazon, Seville
  - Hospital Universitario Río Hortega de Valladolid, Valladolid
- Taiwan (3):
  - Taipei Veterans General Hospital, Taipei
  - TRI-Service General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan

IPD SHARING:
Plan to Share IPD: No